CLINICAL TRIAL: NCT02329119
Title: Psychiatric Disorders and Electrophysiological Markers
Acronym: ERPs-PSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2014-07; RCAPHM14_0077 (Registry Identifier: APHM)
Record Dates: First submitted 2014-12-26; First posted 2014-12-31 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G1-SCZ (Experimental): patients with schizophrenia as defined in DSM IV-TR
  Interventions: Other: electrophysiological recordings
- G2-TAB (Active Comparator): patients with bipolar affective disorder (BD) type I as defined by the DSM IV-TR
  Interventions: Other: electrophysiological recordings

INTERVENTIONS:
Other: electrophysiological recordings

SUMMARY:
Schizophrenia is considered as the most frequent and the most severe chronic psychotic disorder. Its evolutionary modes and its clinical symptomatology remain particularly heterogeneous. Moreover, the brain processes involved in schizophrenia are still far from being clearly understood. Current empirical studies provide a mean duration comprised between 1 and 3 years without any specific diagnosis or treatment. These diagnosis issues are partly based on difficulties in the early distinction between schizophrenia and bipolar affective disorders (BD).

These results emphasize the necessity of new early indices (or endophenotypes). Such markers are intended to be more specific than classical clinical manifestations. In other words, they have to be absent among patients with differential diagnosis, such as BD. Among other possible early indices, several electrophysiological disturbances have been explored.

Our study is designed to mainly describe the N400 component among patients with schizophrenia or BD. This component is classically interpreted as indexing the integration the meaning of a linguistic stimulus in its preceding context. Our main hypothesis aims to show a specific alteration of N400 component among patients with schizophrenia when compared to participants with BD.

The second aim of this study concerns the exploration of four other event related potentials (ERPs) among patients with schizophrenia or BD:

* the P50 component, involved in early sensory gating processes,
* the P300 component, thought to reflect attentional resource allocation and working memory updating of stimulus context,
* the P600 component, elicited during same paradigms than N400, and reflecting their syntactic congruity.
* the CNV (Contingent Negative Variation), reflecting processes of motor anticipation

Regarding to their potential 'endophenotypes' status, our aim consists in comparing the N400 and three other ERPs among patients with schizophrenia or bipolar affective disorder. Since the schizophrenic specificity of such ERPs alterations still remains rarely studied, we also propose to describe the possible relations between these ERPs results and clinical scores observed among patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject showing no severe or progressive somatic pathology, including neurological pathology (head injury, epilepsy, tumor process or multiple sclerosis causing EEG changes incompatible with the observation of ERP characteristics of both psychiatric disorders explored)
* Subject showing a diagnosis of schizophrenia or a diagnosis of bipolar affective disorders, as defined in the DSM IV-TR, in time of inclusion.
* Subject showing no disorder related to the use of a substance according to DSM IV-TR during the last 12 months prior to enrollment.
* Subject not showing another psychiatric disorder according to DSM IV-TR (axis 1 disorders), including schizoaffective disorder or a delusional disorder (not schizophrenic).

Exclusion Criteria:

* Subject unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
amplitude (in µV) of negativity observed the highest between 250 and 500 ms for the N400 component of Event Related Potentials (ERP) | 1 day
  amplitude (in µV) of negativity observed the highest between 250 and 500 ms for the N400 component of Event Related Potentials (ERP) recorded from nine electrodes. For each subject, the average of the amplitude of the nine electrodes is calculated and represents the synthetic parameter for amplitude N400.This is a quantitative parameter. Values will be compared between the two groups of subjects (G1-SCZ and G2-TAB).

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France